CLINICAL TRIAL: NCT04374994
Title: Evaluation of the Clinical and Molecular Efficacy of Daily Avanafil in Egyptian Males With Erectile and Endothelial Dysfunction (Randomized Placebo-Controlled Study)
Brief Title: Daily Avanafil for Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Shimaa Ismail Abdelhamid, MD, Principal investigator, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0105643
Record Dates: First submitted 2020-04-27; First posted 2020-05-05 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; endothelial dysfunction; Avanafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Active Comparator): Males with sexual dysfunction who received daily avanafil tablets (50mg) for four weeks
  Interventions: Drug: Avanafil 50 MG
- control group (Placebo Comparator): Males with sexual dysfunction who received daily placebo tablets for four weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Avanafil 50 MG — Oral phosphodiesterase type 5 inhibitors
  Arms: intervention group
Drug: Placebo oral tablet — lactose and maize starch, Egypt
  Arms: control group

SUMMARY:
In this study, the investigators tried to study the effect of daily avanafil on the serum level of endothelial function markers, as well as its impact on the erectile function in males with erectile and endothelial dysfunction by comparing the results with controls who received placebo.

DETAILED DESCRIPTION:
Avanafil is a highly selective and potent oral phosphodiesterase type 5 inhibitor (PDE5-I) . However, its impact on the soluble markers of endothelial function has not been investigated yet. This study was conducted to assess the effect of daily avanafil on the erectile function and endothelial markers' serum level. In this work we recruited males with erectile dysfunction and other diseases commonly associated with endothelial dysfunction. The investigators randomly treated patients with daily oral avanafil and the other patients with placebo. The investigators measured the International Index of Erectile Function -5 score (IIEF- 5) and the serum levels of markers of endothelial function at baseline and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men with clinical diagnosis of erectile dysfunction of any severity.
* Should be associated with systemic disorders indicative of endothelial dysfunction

Exclusion Criteria:

- Erectile dysfunction due to psychogenic causes, hypogonadism, or spinal cord injury.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
The percentage of change of NO serum level from baseline to 4 weeks | After 4 weeks treatment
  To calculate the percentage of change of Nitric oxide (NO)(in µmol/L) serum level from baseline to 4 weeks post-treatment with avanafil
The percentage of change of cGMP serum level from baseline to 4 weeks | After 4 weeks treatment
  To calculate the percentage of change of cyclic guanosine monophosphate (cGMP) (in pmol/ml) serum level from baseline to 4 weeks post-treatment with avanafil
The percentage of change of ET1 serum level from baseline to 4 weeks | After 4 weeks treatment
  To calculate the percentage of change of endothelin-1 (ET1) (in ng/L) serum level from baseline to 4 weeks post-treatment with avanafil

SECONDARY OUTCOMES:
Comparing avanafil with placebo group regarding post-treatment NO serum levels and percentage of change from baseline. | After 4 weeks treatment
  To compare avanafil with placebo group regarding post-treatment nitric oxide (NO) (in µmol/L) serum level and percentage of change from baseline.
Comparing avanafil with placebo group regarding post-treatment cGMP serum levels and percentage of change from baseline. | After 4 weeks treatment
  To compare avanafil with placebo group regarding posttreatment cyclic guanosine monophosphate (cGMP) (in pmol/ml) serum level and percentage of change from baseline.
Comparing avanafil with placebo group regarding post-treatment ET1 serum levels and percentage of change from baseline. | After 4 weeks treatment
  To compare avanafil with placebo group regarding post-treatment endothelin-1 (ET1) (in ng/L) serum level and percentage of change from baseline.

OTHER OUTCOMES:
Measuring the degree of improvement in the IIEF-5 score | After 4 weeks treatment
  The ED male's clinical response to daily avanafil was subjectively assessed by measuring the degree of improvement in the International Index of Erectile Function scoring (IIEF-5 ) score

CONTACTS AND LOCATIONS:
Overall Officials: Abdelaal Elkamshoushi, MD, Study Director — University of Alexandria
Locations (1):
- Faculty of Medicine, Alexandria University., Alexandria, Elazareta, Egypt

IPD SHARING:
Plan to Share IPD: No
Because we will publish the study in a journal

REFERENCES:
- [Background] Konstantinopoulos A, Giannitsas K, Athanasopoulos A, Spathas D, Perimenis P. The impact of daily sildenafil on levels of soluble molecular markers of endothelial function in plasma in patients with erectile dysfunction. Expert Opin Pharmacother. 2009 Feb;10(2):155-60. doi: 10.1517/14656560802678211. PMID 19236190

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT04374994/Prot_002.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT04374994/SAP_003.pdf